CLINICAL TRIAL: NCT05142345
Title: Randomized Trial of a Care Transition Intervention for Hospitalized Patients With Advanced Cancer
Brief Title: Care Transition Intervention for Hospitalized Patients With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Conquer Cancer Foundation (Other)
Responsible Party: Principal Investigator, Daniel E Lage, MD, MSc, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-501
Record Dates: First submitted 2021-11-20; First posted 2021-12-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Follow-Up Care; Consultation, Remote; Advanced Cancer
Keywords: Cancer; Follow-Up Care; Care Services, Home; Consultation, Remote; Advanced Cancer; Hospitalization; Care Transition Intervention
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTINUUM Intervention Post-Hospital Discharge (Experimental): Participants will receive CONTINUUM intervention visit with a nurse practitioner within three business days of hospital discharge and complete questionnaires about their cancer and care.
  Interventions: Other: CONTINUUM Intervention
- Usual Care Post-Hospital Discharge (Active Comparator): Participants will receive standard oncology care following hospital discharge with follow-up appointments scheduled per primary team and participant preferences. Participants will complete questionnaires about their cancer and care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: CONTINUUM Intervention — The intervention, CONTINUUM (CONTINUity of care Under Management by video visits), consists of a video visit conducted by an oncology nurse practitioner within three business days of hospital discharge, to: (1) reconcile medications, (2) manage symptoms, (3) review the post-hospital care plan for hospitalization-specific issues, and (4) schedule follow-up with the outpatient oncology team.
  Arms: CONTINUUM Intervention Post-Hospital Discharge
Other: Usual Care — Patients assigned to the usual care group will have their post-discharge follow-up scheduled per hospital, outpatient oncology team, and patient preference.
  Arms: Usual Care Post-Hospital Discharge

SUMMARY:
This study is examining whether a care transition intervention, CONTINUUM (CONTINUity of care Under Management by video visits), consisting of a supportive care-focused video visit with an oncology nurse practitioner (NP) within three business days of hospital discharge, may improve post-discharge transitions of care for recently hospitalized patients with advanced cancer.

DETAILED DESCRIPTION:
To address the rising incidence and burden of hospital readmissions for patients with advanced cancer, the investigators developed a population-specific care transition intervention based upon the scholarly literature and our qualitative study. The intervention, CONTINUUM (CONTINUity of care Under Management by video visits), consists of a video visit conducted by an oncology NP within three business days of hospital discharge, to: (1) reconcile medications, (2) manage symptoms, (3) review the post-hospital care plan for hospitalization-specific issues, and (4) schedule follow-up with the outpatient oncology team.

From 01/07/21 to 05/28/21, the investigators conducted a pilot trial of CONTINUUM in 54 patients with advanced cancer recently discharged from the Massachusetts General Hospital Cancer Center (NCT04640714). The investigators found that the intervention was feasible and acceptable in our population.

The investigators are now conducting a randomized controlled trial of the CONTINUUM intervention versus standard of care, to study whether CONTINUUM improves patients' confidence in managing their health condition, as measured by the Patient Activation Measure-13. The investigators will also assess the efficacy of CONTINUUM for improving patient satisfaction with clinician communication, and physical and psychological symptom burden. Lastly, the investigators will explore the effect of the intervention on hospital readmissions within 30-days.

Study procedures include random assignment to either the CONTINUUM intervention or standard oncology care following hospital discharge, questionnaires and medical record data collection.

Participants are expected to be on the study for up to 40 days after hospital discharge.

It is anticipated that about 286 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* First unplanned admission since diagnosis of advanced cancer to to the oncology service at Massachusetts General Hospital (MGH) or the medicine service with oncology consultation
* Known diagnosis of advanced breast, thoracic, genitourinary, gastrointestinal cancers, sarcoma, or melanoma
* Receiving ongoing oncology care at MGH
* Verbal fluency in English
* Internet/wifi or telephone access
* Residing in Massachusetts at the time of hospital discharge

Exclusion Criteria:

* Admitted electively
* Discharged to a location other than home or expired during admission
* Discharged with hospice services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Patients' Confidence in Managing their Health Condition using the Patient Activation Measure-13 (PAM-13) | Baseline to 10-20 days after hospital discharge
  Compare change in the PAM-13 from baseline to 10-20 days post-discharge between study groups. The PAM-13 is scored 0-100 with higher scores indicating greater confidence in managing one's health condition.

SECONDARY OUTCOMES:
Quality of Communication using the Consumer Assessment of Healthcare Providers and Systems (CAHPS) Communication subscale | Up to 10-20 days after hospital discharge
  Compare differences in CAHPS-Communication at up to 10-20 days post-discharge between study groups. CAHPS-Communication has a composite score (score range 0-20) with higher scores indicating better satisfaction. As recommended by CAHPS, we will also analyze specific differences in CAHPS-Communication individual items, which relate to patients' assessment of whether clinicians discussed 1) illness course expectations, 2) what is most important to the patient, and 3) how the treatment plan should match what is most important to the patient. These items are scored as "Yes" vs. "No" responses.
Symptom Burden using the Edmonton Symptom Assessment Scale (ESAS-r) | Baseline to 10-20 days after hospital discharge
  Compare change in the Edmonton Symptom Assessment System-Revised (ESAS-r) total score and physical sub-scale between baseline and 10-20 days of discharge between study groups. Scores on the ESAS-r range from 0-100 with higher scores indicating worse symptom burden. Scores on the ESAS-Physical sub-scale range from 0-70 with higher scores indicating worse symptom burden.
Psychological Symptoms using the Patient Health Questionnaire-4 (PHQ-4) | Baseline to 10-20 days after hospital discharge
  Compare change in the Patient Health Questionnaire-4 (PHQ-4) between baseline and 10-20 days of discharge between study groups. The PHQ-4 is a 4-item tool that contains two 2-item subscales assessing depression and anxiety symptoms. Both subscales and the composite PHQ-4 score can also be evaluated continuously, with higher scores indicating worse psychological distress. Scores on each subscale range from 0 to 6.

OTHER OUTCOMES:
30-day Hospital Readmissions | Up to 30 days after discharge
  Compare hospital readmissions within 30 days of discharge between study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Lage, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation